CLINICAL TRIAL: NCT03258398
Title: A Phase 2, Open-Label, Randomized, Non-Comparative Study With Preliminary Dose Finding to Evaluate eFT508 Monotherapy or eFT508 in Combination With Avelumab in Subjects With Microsatellite Stable Relapsed or Refractory Colorectal Cancer
Brief Title: A Study to Evaluate eFT508 Alone and in Combination With Avelumab in Subjects With MSS Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Effector Therapeutics (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eFT508-0006
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Microsatellite Stable Relapsed or Refractory Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tomivosertib; avelumab

STUDY DESIGN:
Intervention Model Description: In Part 1, subjects will receive eFT508 in combination with a fixed dose of avelumab. Once the recommended dose of eFT508 in combination with avelumab is determined in Part 1, enrollment in Part 2 will begin. Subjects will be randomized in approximately a 2:1 ratio to receive eFT508 in combination with avelumab or eFT508 monotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: eFT508 plus avelumab dose finding Arm (Experimental): subjects will receive eFT508 in combination with a fixed dose of avelumab
  Interventions: Drug: eFT508; Drug: Avelumab
- Part 2: eFT508 plus avelumab (Experimental): subjects will receive eFT508 in combination with a fixed dose of avelumab
  Interventions: Drug: eFT508; Drug: Avelumab
- Part 2: eFT508 alone (Experimental): subjects will receive eFT508 alone
  Interventions: Drug: eFT508

INTERVENTIONS:
Drug: eFT508 — eFT508 will be taken orally (PO) twice a day (bid).
Drug: Avelumab — Avelumab 10 mg/kg will be administered intravenously (IV) on Day 1 and once every 2 weeks (q2wk) thereafter
  Arms: Part 1: eFT508 plus avelumab dose finding Arm; Part 2: eFT508 plus avelumab

SUMMARY:
This is a Phase 2, open-label, 2-part, multicenter study in subjects with MSS relapsed/refractory colorectal cancer. The primary objective of Part 1 is to evaluate the safety and tolerability of escalating doses of eFT508 in combination with a fixed dose of avelumab to determine the maximum tolerated dose (MTD) of eFT508 and to select a recommended dose for Part 2. The primary objective of Part 2 is to evaluate antitumor activity of eFT508 at the recommended dose in combination with avelumab or eFT508 monotherapy. Parts 1 and 2 will also evaluate pharmacokinetics (PK) and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0, 1, or 2
* Pathologically documented diagnosis of colorectal adenocarcinoma.
* Progressed on or intolerant of at least 2 prior cancer therapy regimens administered for metastatic disease.
* Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥3 weeks before the start of study therapy.
* Part 2 only: Presence of radiographically measurable disease (defined as the presence of ≥1 lesion that measures ≥10 mm [≥15 mm for lymph nodes]). Measurable disease that was previously radiated is only permitted if progressing.
* Agrees to undergo a pretreatment and a post-treatment biopsy.
* Microsatellite stable disease determined by IHC and/or polymerase chain reaction (PCR).
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function
* Normal coagulation profile
* Negative antiviral serology
* Female subjects of childbearing potential must not be pregnant or breastfeeding
* Willingness to use protocol-recommended methods of contraception or to abstain from heterosexual intercourse from start of therapy until at lest 30 days after the last dose of study therapy
* Life expectancy of ≥3 months.

Exclusion Criteria:

* History of another malignancy except for adequately treated local basal cell or squamous cell carcinoma of the skin; in situ cervical or breast carcinoma; adequately treated, papillary, noninvasive bladder cancer; other adequately treated Stage 1 or 2 cancers currently in complete remission, or any other cancer that has been in complete remission for ≥2 years.
* Known symptomatic brain metastases requiring ≥10 mg/day of prednisolone (or its equivalent).
* Significant cardiovascular disease.
* Significant screening ECG abnormalities.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Known history of colitis, inflammatory bowel disease, pneumonitis, or pulmonary fibrosis.
* Ongoing risk for bleeding due to active peptic ulcer disease or bleeding diathesis.
* Evidence of an ongoing systemic bacterial, fungal, or viral infection.
* Any condition that may impact the subject's ability to swallow oral medications.
* Major surgery within 4 weeks before the start of study therapy.
* Prior solid organ or bone marrow progenitor cell transplantation.
* Prior therapy with any known inhibitor of MNK-1 or MNK-2.
* Prior therapy with any of the following: PD-1, PD-L1, CTLA4 antibody, or any other drug targeting T cell checkpoint pathways.
* Prior high dose chemotherapy requiring stem cell rescue.
* Intolerance to or prior severe (≥Grade 3) allergic or anaphylactic reaction to infused antibodies or infused therapeutic proteins.
* Vaccination within 4 weeks of the first dose of avelumab and while on study.
* Ongoing immunosuppressive therapy.
* Use of a strong inhibitor or inducer of cytochrome P450 3A4 (CYP3A4) within 7 days prior to the start of study therapy or expected requirement for use of a strong CYP3A4 inhibitor or inducer during study therapy.
* Previously received investigational product in a clinical trial within 30 days or within 5 elimination half lives (whichever is longer) prior to the start of study therapy, or is planning to take part in another clinical trial while participating in this study.
* Has any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, adversely affect the subject's ability to cooperate and participate in the study, or compromise the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Proportion of subjects with a dose limiting toxicity (DLT) during the first treatment cycle | 28 days
Part 2: Overall Response Rate | 8-16 weeks
  the proportion of subjects whose best overall response is a complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Barton, MD, Study Director — CMO
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No